CLINICAL TRIAL: NCT06760468
Title: Functional Probiotic Powder Human Trials
Brief Title: Development and Evaluation of Functional Probiotic Powder in Human Trials
Acronym: FPPHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu Sport University (Other)
Responsible Party: Principal Investigator, Cheng Liang, Director, Chengdu Sport University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SSC202408; 2024YFHZ0077 (Other Grant/Funding Number: Sichuan Provincial Regional Innovation Cooperation Project.)
Record Dates: First submitted 2024-12-26; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Exercise Fatigue
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Randomly select 30 healthy and well-trained athletes aged between 20 and 30 to serve as the experimental group. Participants in the experimental group will undergo an 8-week probiotic powder supplementation intervention. The dosage of the probiotic powder is set at 1x10^9 CFU/kg·bw·d, which means ingesting 10 billion CFU (Colony-Forming Units) of probiotics per kilogram of body weight per day. Before the intervention begins, a comprehensive health assessment and exercise capacity test will be conducted for the participants.
  Blood samples will be collected for baseline biochemical marker analysis. Participants will be instructed to take the probiotic powder once a day at the same time to ensure the consistency of the dosage and the standardization of the intervention.
  Participants will be asked to record their daily consumption, including the time of intake, any omissions, or discomfort. After the 8-week intervention, exercise capacity tests and blood sample collections will be condu
  Interventions: Other: Control; Dietary Supplement: Experimental Group
- Control group (No Intervention): Description: Arm Description: Randomly select 30 healthy and well-trained athletes aged between 20 and 30 to serve as the control group. Participants in the control group will undergo an 8-week placebo supplementation intervention. The placebo has a similar appearance and taste to the probiotic powder but does not contain active probiotic ingredients. Before the intervention begins, a comprehensive health assessment and exercise capacity test will be conducted for the participants. Blood samples will be collected for baseline biochemical marker analysis. Participants will be instructed to take the placebo once a day at the same time to ensure the consistency and standardization of the intervention. Participants will be asked to record their daily consumption, including the time of intake, any omissions, or discomfort. After the 8-week intervention, exercise capacity tests and blood sample collections will be conducted again. Comparing exercise perf

INTERVENTIONS:
Other: Control — Arm Description: Randomly select 30 healthy and well-trained athletes aged between 20 and 30 to serve as the control group. Participants in the control group will undergo an 8-week placebo supplementation intervention. The placebo has a similar appearance and taste to the probiotic powder but does not contain active probiotic ingredients. Before the intervention begins, a comprehensive health assessment and exercise capacity test will be conducted for the participants. Blood samples will be collected for baseline biochemical marker analysis. Participants will be instructed to take the placebo once a day at the same time to ensure the consistency and standardization of the intervention. Participants will be asked to record their daily consumption, including the time of intake, any omissions, or discomfort. After the 8-week intervention, exercise capacity tests and blood sample collections will be conducted again. Comparing exercise performance and biochemical markers before and after t
  Other Names: Control group
  Arms: Experimental group
Dietary Supplement: Experimental Group — Experimental:
  Arm Description: Randomly select 30 healthy and well-trained athletes aged between 20 and 30 to serve as the experimental group. Participants in the experimental group will undergo an 8-week probiotic powder supplementation intervention. The dosage of the probiotic powder is set at 1x10^9 CFU/kg·bw·d, which means ingesting 10 billion CFU (Colony-Forming Units) of probiotics per kilogram of body weight per day. Before the intervention begins, a comprehensive health assessment and exercise capacity test will be conducted for the participants. Blood samples will be collected for baseline biochemical marker analysis. Participants will be instructed to take the probiotic powder once a day at the same time to ensure the consistency of the dosage and the standardization of the intervention. Participants will be asked to record their daily consumption, including the time of intake, any omissions, or discomfort. After the 8-week intervention, exercise ca
  Arms: Experimental group

SUMMARY:
Purpose: To optimize the preparation process of probiotic powder and assess its impact on healthy athletes, providing a scientific basis for functional foods.

Procedures:

Probiotic Powder Preparation: Using vacuum freeze-drying to improve bacterial survival rates.

Human Trials: Recruiting healthy athletes aged 20-30, divided into placebo and probiotic powder groups for an 8-week trial.

Testing and Analysis: Conducting running exhaustion tests and blood biochemical analysis to evaluate the effects of probiotic powder.

Importance: Understanding the effects of probiotics on athletes helps develop better health products.

ELIGIBILITY:
Inclusion Criteria:

* Age Range: Individuals aged 20 to 30 years old.
* Health Status: Healthy, without chronic illnesses or disabilities.
* Athletic Background: Well-trained athletes with a history of regular physical activity.
* Lifestyle: No history of smoking or excessive alcohol consumption.
* Compliance and Consent: Capable of understanding and adhering to study protocols and willing to provide informed consent.

Exclusion Criteria:

* Chronic Illnesses: Individuals with unmanaged chronic diseases
* Substance Use: Current smokers or individuals with a history of substance abuse.
* Allergies and Supplements: History of food allergies or long-term use of nutritional supplements and medications.
* Probiotic and Antibiotic Use: Use of probiotics, fermented products, or antibiotics during the study period.
* Other Conditions: Pregnant or breastfeeding women, individuals with severe mental health conditions, or those participating in other clinical studies.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Lactic acid | 8 weeks
  Lactic acid：Collecting 2 ml of venous blood for measurement indicators
Creatine kinase | 8 weeks
  Creatine kinase: Collecting 2 ml of venous blood for measurement indicators.
Blood urea nitrogen | 8 weeks
  Blood urea nitrogen: Collecting 2 ml of venous blood for measurement indicators.
Liver glycogen | 8 weeks
  Liver glycogen: Collecting 2 ml of venous blood for measurement indicators.
Muscle glycogen | 8 weeks
  Muscle glycogen: Collecting 2 ml of venous blood for measurement indicators.
Total superoxide dismutase | 8 weeks
  Total superoxide dismutase: Collecting 2 ml of venous blood for measurement indicators.
Glutathione | 8 weeks
  Glutathione: Collecting 2 ml of venous blood for measurement indicators.
Malondialdehyde | 8 weeks
  Malondialdehyde

SECONDARY OUTCOMES:
Maximum Oxygen Uptake | 8 weeks
  The cardiopulmonary function testing system provided by the German CORTEX company measures the maximum oxygen uptake.

IPD SHARING:
Plan to Share IPD: No